CLINICAL TRIAL: NCT06714851
Title: Effect of Chondractiv Move (Dietary Supplement) on Activity-related Joint Discomfort in Physically Active Subjects: a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Chondractiv Move on Activity-related Joint Discomfort
Acronym: MOVIPLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Symrise Group (Industry)
Collaborators: CEN Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C1750
Record Dates: First submitted 2024-11-22; First posted 2024-12-04 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Joint; Derangement
Keywords: Activity-related joint discomfort; Collagen hydrolysate

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, single-center study with stratification by gender (~40% men, ~60% women) and menopausal status for women (~50% non-menopausal women, ~50% menopausal women).
  An ancillary subgroup with extended duration of supplementation.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chondractiv Move (Experimental): 8-week supplementation (12 weeks in ancillary subgroup) with 4 capsules/day
  Interventions: Dietary Supplement: Chondractiv Move
- Placebo (Placebo Comparator): 8-week supplementation (12 weeks in ancillary subgroup) with 4 capsules/day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Chondractiv Move — The dietary supplement under study (Chondractiv Move) is a combination of 2 active ingredients: Hydrolyzed chicken cartilage and Rosehip extract at the dose of 1580 mg/day.
  Arms: Chondractiv Move
Other: Placebo — Placebo contains 100% maltodextrins as non-active agent at the dose of 1800 mg/day.
  Arms: Placebo

SUMMARY:
Joint discomfort, manifested as knee pain or gonalgia, is a common problem not only among athletes, but also among people who regularly take part in physical activities and sports. This discomfort can limit mobility and flexibility, even in healthy people who do not suffer from osteoarthritis or other joint diseases. Functional joint discomfort is also due to joint stress and the short-term deterioration of cartilage. The processes of cartilage formation and degradation lose their balance under load, and discomfort is felt for some time after exercise. These conditions and symptoms occur long before the onset of a disease such as osteoarthritis.

Dietary supplements based on herbs or collagen derivatives (a protein involved in maintaining the structure of tissues, including those of the joints) are frequently used to alleviate the discomfort associated with joint disorders and improve the balance between cartilage synthesis and degradation.

This study aims to assess the effect of the dietary supplement "Chondractiv Move" (named "Chondractiv Boost" at the time of protocol writing) on joint discomfort induced by physical activity. This is a combination of rosehip extract and hydrolyzed chicken cartilage containing collagen type II, chondroitin sulfate, and hyaluronic acid as main actives. This combination is chosen based on the results of studies showing the beneficial effects on joints of the ingredients.

DETAILED DESCRIPTION:
This study requires the inclusion of about 140 participants who regularly take part in sporting activities and report knee pain during and/or after this activity.

Participants are randomly assigned to the control group receiving a placebo (a neutral product based on maltodextrins with no effect), or to the test group receiving the dietary supplement. This study is a double-blind, randomized controlled trial. This means that participants as well as assessors do not know the allocation group. This is a necessary procedure to guarantee impartiality in clinical trials.

Participants ingest placebo or dietary supplement for 8 consecutive weeks (or 12 weeks in the ancillary group with extended supplementation duration).

To assess the effect of supplementation, participants are asked to attend medical check-ups and complete questionnaires, before starting the treatment to determine basal values, and then at regular intervals, i.e. every 2 weeks or every month.

Throughout their participation, participants are monitored by the study doctor and must go to a clinical investigation center for doctors visits.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 18.5 and < 30.0 kg/m2.
* Physically active: joint bearing sports (i.e., but not limited to soccer, basketball, handball, volleyball, tennis, running) for at least 3 hours per week or 2 times per week.
* Who self-report activity-related discomfort or reversible knee-joint discomfort during or immediately after physical activity over a period of at least 2 months.
* Who experience pain intensity of 5 (out of 10 on the 11 point-NRS) during the stress joint test (SLSD) and perform at least 25 repetitions.
* Who have no trouble swallowing capsules
* Having a smartphone allowing using the e-PRO App NursTrial®.
* Affiliated to a French Health insurance scheme.
* Signed informed consent.

Exclusion Criteria:

* With diagnosed injury/trauma or tendinopathy (wiper syndrome, patellofemoral syndrome, meniscopathy), algodystrophy, osteoarthritis, rheumatic arthritis or inflammation, or other knee or joint disease.
* Extreme pain symptoms that required high-dose analgesic therapy over a longer period (>2 weeks) or intra-articular injection treatment.
* Untreated or unstable hypothyroidism, or evidence of any neurological disorders.
* Known hypersensitivity to one of the components of the experimental products (i.e., dog rose).
* Intra-articular injections or infiltrations with hyaluronic acid, plasma-rich platelet, glucosamine, chondroitin, or supplementation, with glucosamine, chondroitin, collagen-based products in the last 3 months, or spa therapy related to join health in the last 6 months.
* Current intake of corrective treatment, plant-based products or dietary supplements that could interfere with joint, tendon or bone metabolism.
* May not be compliant or may not respect the constraints imposed by the protocol (i.e., stable physical activities and dietary habits throughout the study).
* Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial.
* For woman of childbearing age (neither menopausal, nor hysterectomised, nor sterilized): not using effective contraception (oral contraceptives, intra-uterine device, contraceptive implant, or condoms).
* Belonging to a population covered by articles L.1121-5 (pregnant confirmed by urinary test at inclusion or breastfeeding women), L.1121-6 (persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care), and L.1121.8 (adults under legal protection or unable to express their consent) of the CSP (French Public Health Code).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline of activity-related joint discomfort at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)
  The pain-related activity is assessed by 0-10 Visual Analogic Scale (VAS) during SLSD (Single-Leg-Step-Down) test.

SECONDARY OUTCOMES:
Change from baseline of activity-related joint discomfort at 4 weeks. | Baseline (Day 0), 4 weeks (Day 28)
  The pain-related activity is assessed by 0-10 Visual Analogic Scale (VAS) during SLSD (Single-Leg-Step-Down) test.
Change from baseline of activity-related joint discomfort at 12 weeks | Baseline (Day 0), 4 weeks (Day 84)
  The pain-related activity is assessed by 0-10 Visual Analogic Scale (VAS) during SLSD (Single-Leg-Step-Down) test.This outcome is only measured in ancillary group.
Activity-related pain at regular exercise/physical activity | Baseline (Day 0), 4 weeks (Day 84)
  Average weekly pain intensity at exercise measured using 0-100 VAS (0 meaning no pain, 100 worst possible pain). At each training session or competition, the subject rates the intensity of pain perceived at exercise.
Change from baseline on overall physical function at 2 weeks | Baseline (Day 0), 2 weeks (Day 14)
  Overall physical function is measured using the Knee injury and Osteoarthritis Outcome Score (KOOS), that consists of 42 items assessing 5 dimensions: pain, other symptoms, activities of daily living, function in sport/recreation, knee related Quality of Life (QoL). KOOS is a self-assessed questionnaire.
Change from baseline on overall physical function at 4 weeks | Baseline (Day 0), 4 weeks (Day 28)
  Overall physical function is measured using the Knee injury and Osteoarthritis Outcome Score (KOOS), that consists of 42 items assessing 5 dimensions: pain, other symptoms, activities of daily living, function in sport/recreation, knee related Quality of Life (QoL). KOOS is a self-assessed questionnaire.
Change from baseline on overall physical function at 6 weeks | Baseline (Day 0), 6 weeks (Day 42)
  Overall physical function is measured using the Knee injury and Osteoarthritis Outcome Score (KOOS), that consists of 42 items assessing 5 dimensions: pain, other symptoms, activities of daily living, function in sport/recreation, knee related Quality of Life (QoL). KOOS is a self-assessed questionnaire.
Change from baseline on overall physical function at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)
  Overall physical function is measured using the Knee injury and Osteoarthritis Outcome Score (KOOS), that consists of 42 items assessing 5 dimensions: pain, other symptoms, activities of daily living, function in sport/recreation, knee related Quality of Life (QoL). KOOS is a self-assessed questionnaire.
Change from baseline on overall physical function at 10 weeks | Baseline (Day 0), 10 weeks (Day 70)
  Overall physical function is measured using the Knee injury and Osteoarthritis Outcome Score (KOOS), that consists of 42 items assessing 5 dimensions: pain, other symptoms, activities of daily living, function in sport/recreation, knee related Quality of Life (QoL). KOOS is a self-assessed questionnaire.
  At week 10, outcome is only measured in ancillary subgroup.
Change from baseline on overall physical function at 12 weeks | Baseline (Day 0), 12 weeks (Day 84)
  Overall physical function is measured using the Knee injury and Osteoarthritis Outcome Score (KOOS), that consists of 42 items assessing 5 dimensions: pain, other symptoms, activities of daily living, function in sport/recreation, knee related Quality of Life (QoL). KOOS is a self-assessed questionnaire.
  At week 12, outcome is only measured in ancillary subgroup.
Change from baseline of knee mobility at 4 weeks | Baseline (Day 0), 4 weeks (Day 28)
  Flexion and extension degrees of the knee measured using the Knee Range of Motion (ROM). Measures is carried out by the investigator using a goniometer.
Change from baseline of knee mobility at 8 weeks | Baseline (Day 0), 8 weeks (D56)
  Flexion and extension degrees of the knee measured using the Knee Range of Motion (ROM). Measures is carried out by the investigator using a goniometer.
Change from baseline of knee mobility at 12 weeks | Baseline (Day 0), 12 weeks (Day 84)
  Flexion and extension degrees of the knee measured using the Knee Range of Motion (ROM). Measures is carried out by the investigator using a goniometer. At week 12, outcome is only measured in ancillary subgroup.
Change from baseline of quality of life at 4 weeks | Baseline (Day 0), 4 weeks (Day 28)
  Quality of life measured using the SF-12, that consists of 12 item-short form of the generic Health-related Quality of Life SF-36. The questionnaire is a self-assessment.
Change from baseline of quality of life at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)
  Quality of life measured using the SF-12, that consists of 12 item-short form of the generic Health-related Quality of Life SF-36. The questionnaire is a self-assessment.
Change from baseline of quality of life at 12 weeks | Baseline (Day 0), 12 weeks (Day 84)
  Quality of life measured using the SF-12, that consists of 12 item-short form of the generic Health-related Quality of Life SF-36. The questionnaire is a self-assessment. At week 12, outcome is only measured in ancillary subgroup.
Satisfaction with the supplementation | 8 weeks (Day 56) or 12 weeks (D84) for ancillary group
  Satisfaction is assessed using a questionnaire with 5-point Likert scale ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) or 4-point Likert scale ((1) Entirely satisfied; (2) Satisfied; (3) Not satisfied; (4) Not satisfied at all), to questions related to the perceived effectiveness.

OTHER OUTCOMES:
Change from baseline of experience of joint pain at 2 weeks | Baseline (Day 0), 2 weeks (Day 14)
  Pain is measured using the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, that consists of 11 items divided into two domains: a 5-item scale for constant pain and a 6-item scale for intermittent pain. ICOAP is a self-assessed questionnaire.
Change from baseline of experience of joint pain at 4 weeks | Baseline (Day 0), 4 weeks (Day 28)
  Pain is measured using the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, that consists of 11 items divided into two domains: a 5-item scale for constant pain and a 6-item scale for intermittent pain. ICOAP is a self-assessed questionnaire.
Change from baseline of experience of joint pain at 6 weeks | Baseline (Day 0), 6 weeks (Day 42)
  Pain is measured using the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, that consists of 11 items divided into two domains: a 5-item scale for constant pain and a 6-item scale for intermittent pain. ICOAP is a self-assessed questionnaire.
Change from baseline of experience of joint pain at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)
  Pain is measured using the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, that consists of 11 items divided into two domains: a 5-item scale for constant pain and a 6-item scale for intermittent pain. ICOAP is a self-assessed questionnaire.
Change from baseline of experience of joint pain at 10 weeks | Baseline (Day 0), 10 weeks (Day 70)]
  Pain is measured using the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, that consists of 11 items divided into two domains: a 5-item scale for constant pain and a 6-item scale for intermittent pain. ICOAP is a self-assessed questionnaire. At week 10, outcome is only measured in ancillary subgroup.
Change from baseline of experience of joint pain at 12 weeks | Baseline (Day 0), 12 weeks (Day 84)
  Pain is measured using the Intermittent and Constant Osteoarthritis Pain (ICOAP) questionnaire, that consists of 11 items divided into two domains: a 5-item scale for constant pain and a 6-item scale for intermittent pain. ICOAP is a self-assessed questionnaire. At week 12, outcome is only measured in ancillary subgroup.
Change from baseline in cartilage synthesis at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)
  Serum concentrations of Type IIA collagen N-propeptide are measured using ELISA assays.
Change from baseline in cartilage degradation at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)]
  Serum concentrations of Cartilage oligomeric matrix protein (COMP) are measured using ELISA assays.
Impression improvement of joint function/discomfort at 2 weeks | Baseline (Day 0), 2 weeks (Day 14)
  Subjective impression of improvement is self-assessed by the subject using a 5-point Likert scale: ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) in response to "Since I started the supplementation, I am feeling an improvement: of my knee mobility/ knee stiffness/ joint comfort during physical activity/ joint comfort during daily activities".
Impression improvement of joint function/discomfort at 4 weeks | Baseline (Day 0), 4 weeks (Day 28)
  Subjective impression of improvement is self-assessed by the subject using a 5-point Likert scale: ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) in response to "Since I started the supplementation, I am feeling an improvement: of my knee mobility/ knee stiffness/ joint comfort during physical activity/ joint comfort during daily activities".
Impression improvement of joint function/discomfort at 6 weeks | Baseline (Day 0), 6 weeks (Day 42)
  Subjective impression of improvement is self-assessed by the subject using a 5-point Likert scale: ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) in response to "Since I started the supplementation, I am feeling an improvement: of my knee mobility/ knee stiffness/ joint comfort during physical activity/ joint comfort during daily activities".
Impression improvement of joint function/discomfort at 8 weeks | Baseline (Day 0), 8 weeks (Day 56)
  Subjective impression of improvement is self-assessed by the subject using a 5-point Likert scale: ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) in response to "Since I started the supplementation, I am feeling an improvement: of my knee mobility/ knee stiffness/ joint comfort during physical activity/ joint comfort during daily activities".
Impression improvement of joint function/discomfort at 10 weeks | Baseline (Day 0), 10 weeks (Day 70)
  Subjective impression of improvement is self-assessed by the subject using a 5-point Likert scale: ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) in response to "Since I started the supplementation, I am feeling an improvement: of my knee mobility/ knee stiffness/ joint comfort during physical activity/ joint comfort during daily activities". At week 10, outcome is only measured in ancillary subgroup.
Impression improvement of joint function/discomfort at 12 weeks | Baseline (Day 0), 12 weeks (Day 84)
  Subjective impression of improvement is self-assessed by the subject using a 5-point Likert scale: ((1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree)) in response to "Since I started the supplementation, I am feeling an improvement: of my knee mobility/ knee stiffness/ joint comfort during physical activity/ joint comfort during daily activities". At week 12, outcome is only measured in ancillary subgroup.
Evaluation of therapeutic saving | 8 weeks (Day 56) or 12 weeks (Day 84) in ancillary subgroup
  Consumption of anti-inflammatory and analgesic drugs taken to relieve knee pain (name, number, dose) and recorded by the subject from Day 0 to Day 56, and Day 0 to Day 84 in ancillary subgroup. Drug consumption is expressed as equivalent doses of ibuprofen or paracetamol.
Adverse effect | 8 weeks (Day 56) or 12 weeks (Day 84) in ancillary subgroup
  Adverse events are described using the MedDRA dictionary. Adverse event with possible relation to the experimental products are classified by type of adverse reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Christine JUHEL, Ph.D, Study Chair — CEN Biotech; Carole PERRIN, MD, Principal Investigator — CEN Biotech
Locations (1):
- Cen Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No
Subjects data is not anonymized. To comply with European regulations and national provisions, subjects are informed that no sharing of IPD is planned in order to protect their personal data. If data is to be shared, patients must be informed individually, and their consent obtained.
  At this stage, only aggregated data can be shared